CLINICAL TRIAL: NCT00394966
Title: A Phase 2, MultiCenter, Randomized, Placebo-Controlled, Double-Blind, Dose Finding Study to Determine the Safety and Efficacy of SCH 619734 for the Treatment of Chemotherapy Induced Nausea and Vomiting (CINV) in Subjects Receiving Highly Emetogenic Chemotherapy (HEC)
Brief Title: A Multicenter, Randomized, Controlled Trial of SCH 619734 for the Treatment of Chemotherapy-Induced Nausea and Vomiting (Study P04351AM2)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P04351; Study ID: 3283299
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — rolapitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- SCH 619734 Dose 1 (Experimental)
  Interventions: Drug: SCH 619734 Dose 1
- SCH 619734 Dose 2 (Experimental)
  Interventions: Drug: SCH 619734 Dose 2
- SCH 619734 Dose 3 (Experimental)
  Interventions: Drug: SCH 619734 Dose 3
- SCH 619734 Dose 4 (Experimental)
  Interventions: Drug: SCH 619734 Dose 4
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCH 619734 Dose 1 — SCH 619734 10 mg (4 capsules) x 1 orally approximately 2 hours prior to the administration of the first chemotherapeutic agent on Day 1 of Cycle 1 and on Day 1 of all subsequent cycles (up to five additional cycles)
  Other Names: Rolapitant
  Arms: SCH 619734 Dose 1
Drug: SCH 619734 Dose 2 — SCH 619734 25 mg (4 capsules) x 1 orally approximately 2 hours prior to the administration of the first chemotherapeutic agent on Day 1 of Cycle 1 and on Day 1 of all subsequent cycles (up to five additional cycles)
  Other Names: Rolapitant
  Arms: SCH 619734 Dose 2
Drug: SCH 619734 Dose 3 — SCH 619734 100 mg (2 capsules) x 1 orally approximately 2 hours prior to the administration of the first chemotherapeutic agent on Day 1 of Cycle 1 and on Day 1 of all subsequent cycles (up to five additional cycles)
  Other Names: Rolapitant
  Arms: SCH 619734 Dose 3
Drug: SCH 619734 Dose 4 — SCH 619734 200 mg (4 capsules) x 1 orally approximately 2 hours prior to the administration of the first chemotherapeutic agent on Day 1 of Cycle 1 and on Day 1 of all subsequent cycles (up to five additional cycles)
  Other Names: Rolapitant
  Arms: SCH 619734 Dose 4
Drug: Placebo — Matching placebo x 1 orally approximately 2 hours prior to the administration of the first chemotherapeutic agent on Day 1 of Cycle 1 and on Day 1 of all subsequent cycles (up to five additional cycles)
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, multicenter, parallel-group, double-blind, placebo-controlled study of various doses of SCH 619734 in subjects receiving cisplatin-based chemotherapy. Ondansetron and dexamethasone will be concurrently administered with SCH 619734 before initiation of chemotherapy on Day 1. Subjects will record nausea and vomiting in the SPNV Subject Diary through Day 6. The quality of life assessment as measured by the Functional Living Index-Emesis Questionnaire (FLIE) will be used to measure the effect of chemotherapy-induced nausea and vomiting (CINV) on daily life. Blood samples for SCH 619734 pharmacokinetic assessments will be collected. The study is to be conducted in conformance with Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject has never been treated with cisplatin and is to receive first course of cisplatin-based chemotherapy (>=70 mg/m^2).
* Subject has a Karnofsky performance score of >=60.
* Subject has a predicted life expectancy of >=3 months.
* Subject has adequate bone marrow, kidney, and liver function as evidenced by:

  * Absolute neutrophil count >=1,500/mm3 and white blood cell count >=3,000/mm3.
  * Platelet count >=100,000/mm3.
  * Aspartate aminotransferase (AST) <=2.5 x upper limit of normal (ULN) range.
  * Alanine aminotransferase (ALT) <=2.5 x ULN.
  * Bilirubin <=1.5 x ULN, except for subjects with Gilbert's syndrome.
  * Creatinine <=1.5 x ULN.
* Subject is able to read, understand, and complete the questionnaires.

Exclusion Criteria:

* Any current treatment or medical history (eg, subject is mentally incapacitated or has a psychiatric disorder) that, in the opinion of the investigator, would confound the results of the study or pose any unwarranted risk in administering study drug to the subject.
* Subject has contraindication to the administration of cisplatin, ondansetron, or dexamethasone including, but not limited to, a history of hypersensitivity to the drugs or their components, severe renal impairment, severe bone marrow suppression, hearing impairment, or systemic fungal infection.
* Subject is scheduled to receive any other chemotherapeutic agent with an emetogenicity level of 3 or above (Hesketh Scale) from Day -2 through Day 6.
* Subject is scheduled to receive any radiation therapy to the abdomen or pelvis within 5 days prior to and/or during Days 1 through 5 following cisplatin infusion.
* Subject has symptomatic primary or metastatic central nervous system (CNS) disease.
* Subject has ongoing vomiting caused by any etiology or has a history of anticipatory nausea and vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the overall complete response rate (no emesis and no use of rescue medication from 0 through 120 hours following initiation of cisplatin-based chemotherapy). | Days 1 through 6.

SECONDARY OUTCOMES:
The key secondary efficacy endpoints are the complete response rates for the acute (0 through 24 hours) and delayed (>24 through 120 hours) phases of CINV. | Days 1 through 6.
The key secondary safety endpoints are adverse events, physical examinations, vital signs, electrocardiograms, and safety laboratory values. | Throughout the study and up to 30 days after the subject completes or discontinues from the study.